CLINICAL TRIAL: NCT03019380
Title: Testing the Effectivness and Safety of the Wondertip
Brief Title: A Clinical Trial to Test the Saftey and Success Rate for a Cerrumen Cleaning Device - "Wondertip".
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Dr Udi Katzanel, head of otology and cochlear implant program, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0125-16-KMC-CTIL
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: External Ear Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Impacted cerumen (Experimental): removing cerumen from external ears of patients with impacted cerumen, obscuring the canal and the tympanic membrane.
  Interventions: Device: removing cerumen from external ear (Wondertip)

INTERVENTIONS:
Device: removing cerumen from external ear (Wondertip) — The wondertip will be coiled into the external ear canal with the purpose of grasping and evacuating the cerumen. Following the evacuation, the depth of the external ear canal will be messured.

SUMMARY:
Wondertip is a silicone single use device with a coil end, designed for the purpose of evacuating impacted cerumen of external ear canals. This trial aims at testing the safety and efficacy of this device. The participating investigators will be ENT doctors with the skill of examining the treating ear problems.

DETAILED DESCRIPTION:
Cerumen is ear wax, a combination of dead skin cells of the external ear canal, sebaceous glands secretions and ceruminous sweat glands secretions. Cerumen exists in a range of people but sometimes it become an obstacle to patients or caregivers. Cerumen may accumulate in the external ear canal and cause discomfort to the patient, sensation ofobtuseness and conductive hearing loss. Patients who use hearing aids may suffer from problems wearing them, and sometimes the cerumen may plug the inner part of the hearing aid or the ventilation channel of the ear phone.

For caregivers, cerumen may poses a diagnostic challenge, by concealing part of the external ear canal and tympanic membrane, thus making it difficult to observe the middle ear. cerumen my affect the results of audiometric tests, ABR tests, Otoacustic Emission tests and in conducting tympanometric tests. All of which may result in false results. The incidence of cerumen is estimated to be betwean 7 to 35% of the general population.

There are few options to evacuate the cerumen, but they usually require skill and the use of otology microscope. It mays casue discomfort or pain, and even trauma to the external ear canal or the tympanic membrane. A device which does not require a special skill or equipment may have a advantage, especially for the general practioner doctor.

The Wondertip is an Israeli patent, made of silicone with a coil like end, targeted to evacuate the cerumen in a safe and effective manner. The coil is gently inserted to the ear canal, grasps and evacuates the cerumen.

The purpose of the trial is to investigate the safety and efficacy of the Wondertip. A second purpose is to messure external ear canal depth.

Each candidate which will present with cerumen impaction will recieve a detailed explanation regarding the trial. If the patient agrees, and signs a concent form, a short interview will take place by the doctor. An evacuation of the cerumen will be attempted by the same doctor with the Wondertip. Further the doctor will document details regarding the safety and efficacy of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 1 year old who have cerumen impaction.

Exclusion Criteria:

* external ear infection
* chronic otitis media with perforation of the tympanic membrane
* past ear surgery
* otorrhea
* inflamation of the auricle or the periauricular region
* temporal bone neoplasm
* deafness in the contralateral ear (single sided deafness).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
view of the tympanic membrane | 10 minutes
  how much of the tympanic is visible after using the Wondertip

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Katzanel, Dr, Principal Investigator — Kaplan Medical Center

IPD SHARING:
Plan to Share IPD: No
no plan of sharing IPD